CLINICAL TRIAL: NCT04954625
Title: Prolonged Air Leak (PAL) Autologous Blood Patch Intervention Trial
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Rush University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 19072606
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Lung Cancer
Keywords: Surgery; Prolonged Air Leak; Autologous Blood Patch; Lung
MeSH Terms: conditions — Lung Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autologous Blood Patch (Experimental): 60-120ml of patient's blood will be drawn and inserted into patient's chest tube. A minimum of 60ml of blood is required, with the optimal amount of blood being 120ml.
  Interventions: Procedure: Autologous Blood Patch
- Standard of Care (Per physician) (Active Comparator): Chest tube remains intact without blood patch.
  Interventions: Procedure: Standard of Care (per Physician)

INTERVENTIONS:
Procedure: Autologous Blood Patch — All patients will be assessed on the morning of postoperative Day 3 and 4 for the presence of an air leak. If an air leak is present, 60-100 ml of autologous blood will be drawn from a peripheral vein and immediately instilled into the chest tube. The individual who draws blood is that the discretion of the site principal investigator. The tubing will be elevated over an IV pole while the patient remains in bed, moving position every 15 minutes for 1 hour to distribute the blood throughout the pleural cavity. The tubing support will then be removed, allowing the chest tube to drain. After ABP intervention, the chest tube will remain to water seal, as long as the patient tolerates it.
  Arms: Autologous Blood Patch
Procedure: Standard of Care (per Physician) — Patients randomized to Standard of Care will be treated as their surgeon would as routine. This may mean postoperative observation, of another type of intervention.
  Arms: Standard of Care (Per physician)

SUMMARY:
A postoperative autologous blood patch (ABP) intervention trial for patients who underwent lung resection for cancer to examine its effectiveness in preventing a prolonged air leak.

AIM 1: To determine the safety and efficacy of autologous blood patch (ABP) as a means to reduce the rate of prolonged air leak (PAL) after lung cancer resection

AIM 2: To prospectively examine variation in morbidity and quality of life between patients with and without a PAL

DETAILED DESCRIPTION:
The plan for this trial is to establish the safety and efficacy of ABP as a means of reducing PAL following lung cancer resection. Patients with an air leak on the morning of postoperative day 3 after elective lung resection for cancer will be randomized to ABP on postoperative day 3 and day 4 (if an air leak remains present), or standard care (n=60 per arm). This will be a multi-institutional randomized, controlled trial open for enrollment at centers in the United States and Canada. The study methods and design are compliant with the Consolidated Standards of Reporting Trials (CONSORT).

Subjects will be consented on postoperative day 3, with autologous blood patch intervention occurring on day 3 or day 4. If subjects are randomized to the ABP arm of the trial, they will receive 60-100 ml of autologous blood sterilely drawn from a peripheral vein and immediately instilled into the chest tube.

Subjects will then follow up either in clinic or via telephone to answer the questionnaire. If the subject is being seen in person, they will be handed a questionnaire form to complete. This form will be kept and stored as source documentation. If the patient is answering the questionnaire via telephone, the study team personnel will record their answers on the questionnaire form, indicating it was completed by the subject but recorded by study team personnel. A telephone encounter note will be recorded and stored as source with the completed questionnaire. Follow up occurs at 30 days (+/-5 days) postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent elective wedge resection, segmentectomy, lobectomy, or bilobectomy for suspected non-small cell lung cancer
* Patients that have reviewed and signed the Informed Consent Form, had an opportunity to ask questions, and consent to have their de-identified data included in the study
* Patients who have an air leak on the morning of postoperative Day 3
* Age ≥18 years old

Exclusion Criteria:

* Patients who undergo pneumonectomy, sleeve lobectomy, chest wall or diaphragm resection, or bilateral procedures.
* Age < 18 years old
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prolonged Air Leak >5 days | Within 30 Days
  Definition of prolonged air leak: air leak present at 5 days or greater
Hospital Length of Stay | Within 30 Days
  Number of days patient was admitted inpatient
Readmission within 30 days | Within 30 Days
  Determination of whether the patient was readmitted after discharge within 30 days.
In hospital mortality | Within 30 Days
  Survival status while inpatient.
30-day Mortality | Within 30 Days
  Survival status within 30 days consent.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Seder, MD, Principal Investigator — Rush University Medical Center; Sebastien Gilbert, MD, Study Director — University of Ottawa
Locations (1):
- Rush University Medical Center, Chicago, Illinois, United States

REFERENCES:
- [Background] U.S. Cancer Statistics Working Group. United States Cancer Statistics: 1999-2013 Incidence and Mortality Web-based Report. Atlanta: U.S. Department of Health and Human Services, Centers for Disease Control and Prevention and National Cancer Institute; 2017. Available at: www.cdc.gov/uscs
- [Background] Stephan F, Boucheseiche S, Hollande J, Flahault A, Cheffi A, Bazelly B, Bonnet F. Pulmonary complications following lung resection: a comprehensive analysis of incidence and possible risk factors. Chest. 2000 Nov;118(5):1263-70. doi: 10.1378/chest.118.5.1263. PMID 11083673
- [Background] Brunelli A, Monteverde M, Borri A, Salati M, Marasco RD, Fianchini A. Predictors of prolonged air leak after pulmonary lobectomy. Ann Thorac Surg. 2004 Apr;77(4):1205-10; discussion 1210. doi: 10.1016/j.athoracsur.2003.10.082. PMID 15063235
- [Background] Isowa N, Hasegawa S, Bando T, Wada H. Preoperative risk factors for prolonged air leak following lobectomy or segmentectomy for primary lung cancer. Eur J Cardiothorac Surg. 2002 May;21(5):951. doi: 10.1016/s1010-7940(02)00076-3. No abstract available. PMID 12062302
- [Background] Liang S, Ivanovic J, Gilbert S, Maziak DE, Shamji FM, Sundaresan RS, Seely AJE. Quantifying the incidence and impact of postoperative prolonged alveolar air leak after pulmonary resection. J Thorac Cardiovasc Surg. 2013 Apr;145(4):948-954. doi: 10.1016/j.jtcvs.2012.08.044. Epub 2012 Sep 13. PMID 22982031
- [Background] Gilbert S, Maghera S, Seely AJ, Maziak DE, Shamji FM, Sundaresan SR, Villeneuve PJ. Identifying Patients at Higher Risk of Prolonged Air Leak After Lung Resection. Ann Thorac Surg. 2016 Nov;102(5):1674-1679. doi: 10.1016/j.athoracsur.2016.05.035. Epub 2016 Jul 22. PMID 27457828
- [Background] Attaar A, Winger DG, Luketich JD, Schuchert MJ, Sarkaria IS, Christie NA, Nason KS. A clinical prediction model for prolonged air leak after pulmonary resection. J Thorac Cardiovasc Surg. 2017 Mar;153(3):690-699.e2. doi: 10.1016/j.jtcvs.2016.10.003. Epub 2016 Oct 14. PMID 27912898
- [Background] Lee L, Hanley SC, Robineau C, Sirois C, Mulder DS, Ferri LE. Estimating the risk of prolonged air leak after pulmonary resection using a simple scoring system. J Am Coll Surg. 2011 Jun;212(6):1027-32. doi: 10.1016/j.jamcollsurg.2011.03.010. Epub 2011 Apr 13. PMID 21489831
- [Background] Brunelli A, Varela G, Refai M, Jimenez MF, Pompili C, Sabbatini A, Aranda JL. A scoring system to predict the risk of prolonged air leak after lobectomy. Ann Thorac Surg. 2010 Jul;90(1):204-9. doi: 10.1016/j.athoracsur.2010.02.054. PMID 20609776
- [Background] Rivera C, Bernard A, Falcoz PE, Thomas P, Schmidt A, Benard S, Vicaut E, Dahan M. Characterization and prediction of prolonged air leak after pulmonary resection: a nationwide study setting up the index of prolonged air leak. Ann Thorac Surg. 2011 Sep;92(3):1062-8; discussion 1068. doi: 10.1016/j.athoracsur.2011.04.033. PMID 21871301
- [Background] Stolz AJ, Schutzner J, Lischke R, Simonek J, Pafko P. Predictors of prolonged air leak following pulmonary lobectomy. Eur J Cardiothorac Surg. 2005 Feb;27(2):334-6. doi: 10.1016/j.ejcts.2004.11.004. PMID 15691692
- [Background] Pompili C, Falcoz PE, Salati M, Szanto Z, Brunelli A. A risk score to predict the incidence of prolonged air leak after video-assisted thoracoscopic lobectomy: An analysis from the European Society of Thoracic Surgeons database. J Thorac Cardiovasc Surg. 2017 Apr;153(4):957-965. doi: 10.1016/j.jtcvs.2016.11.064. Epub 2016 Dec 22. PMID 28089646
- [Background] Varela G, Jimenez MF, Novoa N, Aranda JL. Estimating hospital costs attributable to prolonged air leak in pulmonary lobectomy. Eur J Cardiothorac Surg. 2005 Feb;27(2):329-33. doi: 10.1016/j.ejcts.2004.11.005. PMID 15691691
- [Background] Liberman M, Muzikansky A, Wright CD, Wain JC, Donahue DM, Allan JS, Gaissert HA, Morse CR, Mathisen DJ, Lanuti M. Incidence and risk factors of persistent air leak after major pulmonary resection and use of chemical pleurodesis. Ann Thorac Surg. 2010 Mar;89(3):891-7; discussion 897-8. doi: 10.1016/j.athoracsur.2009.12.012. PMID 20172150
- [Background] Mueller MR, Marzluf BA. The anticipation and management of air leaks and residual spaces post lung resection. J Thorac Dis. 2014 Mar;6(3):271-84. doi: 10.3978/j.issn.2072-1439.2013.11.29. PMID 24624291
- [Background] Okereke I, Murthy SC, Alster JM, Blackstone EH, Rice TW. Characterization and importance of air leak after lobectomy. Ann Thorac Surg. 2005 Apr;79(4):1167-73. doi: 10.1016/j.athoracsur.2004.08.069. PMID 15797045
- [Background] Elsayed H, McShane J, Shackcloth M. Air leaks following pulmonary resection for lung cancer: is it a patient or surgeon related problem? Ann R Coll Surg Engl. 2012 Sep;94(6):422-7. doi: 10.1308/003588412X13171221592258. PMID 22943333
- [Background] Seder CW, Basu S, Ramsay T, Rocco G, Blackmon S, Liptay MJ, Gilbert S. A Prolonged Air Leak Score for Lung Cancer Resection: An Analysis of The Society of Thoracic Surgeons General Thoracic Surgery Database. Ann Thorac Surg. 2019 Nov;108(5):1478-1483. doi: 10.1016/j.athoracsur.2019.05.069. Epub 2019 Jul 16. PMID 31323209
- [Background] Rocco G, Brunelli A, Rocco R. Suction or Nonsuction: How to Manage a Chest Tube After Pulmonary Resection. Thorac Surg Clin. 2017 Feb;27(1):35-40. doi: 10.1016/j.thorsurg.2016.08.006. PMID 27865325
- [Background] Rivas de Andres JJ, Blanco S, de la Torre M. Postsurgical pleurodesis with autologous blood in patients with persistent air leak. Ann Thorac Surg. 2000 Jul;70(1):270-2. doi: 10.1016/s0003-4975(00)01360-6. PMID 10921721
- [Background] Lang-Lazdunski L, Coonar AS. A prospective study of autologous 'blood patch' pleurodesis for persistent air leak after pulmonary resection. Eur J Cardiothorac Surg. 2004 Nov;26(5):897-900. doi: 10.1016/j.ejcts.2004.07.034. PMID 15519179
- [Background] Oliveira FH, Cataneo DC, Ruiz RL Jr, Cataneo AJ. Persistent pleuropulmonary air leak treated with autologous blood: results from a university hospital and review of literature. Respiration. 2010;79(4):302-6. doi: 10.1159/000226277. Epub 2009 Jun 24. PMID 19556743
- [Background] Athanassiadi K, Bagaev E, Haverich A. Autologous blood pleurodesis for persistent air leak. Thorac Cardiovasc Surg. 2009 Dec;57(8):476-9. doi: 10.1055/s-0029-1185913. PMID 20013622
- [Background] Shackcloth MJ, Poullis M, Jackson M, Soorae A, Page RD. Intrapleural instillation of autologous blood in the treatment of prolonged air leak after lobectomy: a prospective randomized controlled trial. Ann Thorac Surg. 2006 Sep;82(3):1052-6. doi: 10.1016/j.athoracsur.2006.04.015. PMID 16928534
- [Background] Chambers A, Routledge T, Bille A, Scarci M. Is blood pleurodesis effective for determining the cessation of persistent air leak? Interact Cardiovasc Thorac Surg. 2010 Oct;11(4):468-72. doi: 10.1510/icvts.2010.234559. Epub 2010 Jul 13. PMID 20628018
- [Background] Manley K, Coonar A, Wells F, Scarci M. Blood patch for persistent air leak: a review of the current literature. Curr Opin Pulm Med. 2012 Jul;18(4):333-8. doi: 10.1097/MCP.0b013e32835358ca. PMID 22498731
- [Background] Cobanoglu U, Melek M, Edirne Y. Autologous blood pleurodesis: A good choice in patients with persistent air leak. Ann Thorac Med. 2009 Oct;4(4):182-6. doi: 10.4103/1817-1737.56011. PMID 19881163
- [Background] Cagirici U, Sahin B, Cakan A, Kayabas H, Buduneli T. Autologous blood patch pleurodesis in spontaneous pneumothorax with persistent air leak. Scand Cardiovasc J. 1998;32(2):75-8. doi: 10.1080/14017439850140210. PMID 9636962
- [Background] Viale PH. The American Cancer Society's Facts & Figures: 2020 Edition. J Adv Pract Oncol. 2020 Mar;11(2):135-136. doi: 10.6004/jadpro.2020.11.2.1. Epub 2020 Mar 1. No abstract available. PMID 33532112
- [Background] National Lung Screening Trial Research Team; Aberle DR, Adams AM, Berg CD, Black WC, Clapp JD, Fagerstrom RM, Gareen IF, Gatsonis C, Marcus PM, Sicks JD. Reduced lung-cancer mortality with low-dose computed tomographic screening. N Engl J Med. 2011 Aug 4;365(5):395-409. doi: 10.1056/NEJMoa1102873. Epub 2011 Jun 29. PMID 21714641